CLINICAL TRIAL: NCT01841866
Title: Does Laryngeal Mask Airway Removal During Deep Anesthesia Reduce Postoperative Sore Throat in Children?
Brief Title: Laryngeal Mask Airway Removal During Deep Anesthesia in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Ngamjit Pattaravit, Doctor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LMA246521
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Post Operative Sore Throat After LMA Removal
Keywords: post operative sore throat; laryngeal mask airway; children

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- deep anesthetic state (Active Comparator): LMA removal
  Interventions: Other: LMA removal
- awake (Placebo Comparator): LMA removal
  Interventions: Other: LMA removal

INTERVENTIONS:
Other: LMA removal

SUMMARY:
Laryngeal mask airway (LMA) is widely used in children.The appropriate time to remove laryngeal mask airway is still inconclusive.Sore throat is one of common complications after general anesthesia. Sometimes postoperative sore throat affects patients' satisfaction and daily activities. It can be correlated with dysphagia and may limit oral intake especially in children.The incidence of postoperative sore throat after laryngeal mask airway insertion varies from 5.8-34% in adult(13) and 17.5% in pediatric.Somehow, almost the studies of postoperative sore throat after laryngeal mask airway removal were done in awake state. Our study object to test that post operative sore throat after LMA removal in deep anesthetized children is lower than awake children.

DETAILED DESCRIPTION:
Patients age between 6-12 years who have ASA physical status I-II and scheduled for elective surgery will be enrolled in this study and randomly assigned into two groups (group A = awake group and group D = deep anesthetized group) by using computer-generated randomization table. The patients who have the following problems: active airway disease, risk of aspiration, intra-peritoneal or airway surgery will be excluded.

At the day of surgery, demographic data will be recorded by nurse anesthetist. Visual analog scale (VAS) will be used as a tool for evaluating preoperative sore throat.

At the operating room, after standard monitoring and pre-oxygenated with 100% oxygen via tight anesthetic face mask for 5 minutes. Propofol (3-5 mg/kg) and fentanyl(1-3 ug/kg) will be used for induction. After the patient is apnea and loss of eyelash reflex, appropriate size of classic LMA ,which is prepared by fully deflated to forms a smooth "spoon-shape" and be lubricated by water based jelly, will be applied with standard LMA insertion technique. Once LMA is in the right position, air will be inflated to the cuff of LMA, for keeping cuff pressure between 40-60 cmH2O. Air, O2 and Sevoflurane ≥ 1minimal alveolar concentration (MAC) will be used to keep the patient anesthetized. Performer of LMA insertion and number of insertion attempts will be recorded.

At the end of surgery, LMA will be removed with the technique which is followed by the group assignment, group D and group A. After that, patient will be transferred to post anesthetic care unit (PACU).

At PACU, After the patient is fully awake, the blind investigator will ask the patient to evaluate post operative sorethroat by using Visual analog scale (VAS) (0-10). Dysphagia (discomfort when swallowing) using dysphagia score (0 = able to eat normal diet / no dysphagia, 1 = able to swallow some solid foods, 2 = able to swallow only semi solid foods, 3 = able to swallow liquids only, 4 = unable to swallow anything / total dysphagia), dysphonia (discomfort when speaking such as hoarseness) using dysphonia score (0 = no hoarseness, 1 = mild/no hoarseness in the time of interview but had it previously, 2 = moderate/only is felt by the patient or their parents, 3 = severe/recognizable in the time of interview) Any adverse events will be evaluated at 1 hour in PACU. Then the evaluation will be repeated by telephoned interview at 24 and 72 hours respectively.

ELIGIBILITY:
Inclusion Criteria:

* age 6-12 years
* ASA physical status I-II
* elective surgery

Exclusion Criteria:

* active airway disease
* risk for aspiration
* intraperitoneal or airway surgery

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 456 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Sorethroat | upto 72 hr post operative period
  Evaluate post operative sorethroat by using Visual analog scale (VAS) (0-10)

SECONDARY OUTCOMES:
Dysphagia | upto 72 hr postoperative period
  Dysphagia (discomfort when swallowing) by using Visual analog scale (VAS) (0-10) dysphagia score 0 = able to eat normal diet / no dysphagia
  1. = able to swallow some solid foods
  2. = able to swallow only semi solid foods
  3. = able to swallow liquids only
  4. = unable to swallow anything / total dysphagia
Dysphonia | upto 72 hr postoperative period
  dysphonia (discomfort when speaking such as hoarseness) by using numerical rating scale (VAS) (0-10) dysphonia score 0= no hoarseness
  1. = mild/no hoarseness in the time of interview but had it previously
  2. = moderate/only is felt by the patient or their parents
  3. = severe/recognizable in the time of interview
Adverse event: teeth or mucosal trauma | upto 72 hr postoperative period
  Yes /no
laryngospasm | Intraoperative and PACU period
  yes/ no
Bronchospasm | Intraoperative and PACU period
  yes/no
Desaturation | Intraoperative and PACU period
  Oxygen saturation less than 95%
Nausea and vomiting | up to 72 hr postoperative period
  using numerical rating scale (VAS) (0-10) as a measurement tool
cough | up to72 hr postoperative period
  Mild: < 10 times per day Moderate 10-20 times per day Severe > 20 times per day

CONTACTS AND LOCATIONS:
Overall Officials: Ngamjit Pattaravit, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand